CLINICAL TRIAL: NCT02956265
Title: Assessment of Optical Spectroscopy's Diagnosis Accuracy When Non-invasively and Automatically Classifying Skin Lesions in One of the Following Histological Classes: Healthy, Actinic Keratosis, in Situ Carcinoma and Invasive Carcinoma.
Brief Title: Optical Spectroscopy for Skin Carcinomas' Surgical Management
Acronym: SPECTROLIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-05-CHRMT
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2021-06

CONDITIONS: Carcinomatous or Polymorphous Skin Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients - Suffering from carcinomatous or polymorphous skin (Experimental)
  Interventions: Device: bimodal optical spectroscopy

INTERVENTIONS:
Device: bimodal optical spectroscopy — an optical fiber will be put in gentle contact with the patient's skin in order to acquire optical spectra

SUMMARY:
Actinic keratosis are of utmost medical and economical interest because of their high prevalence (20 % of 60 year-old people and older in the Northern hemisphere) and their important cosmetic impact as such actinic keratosis mostly appear on photo-exposed skin sites. The surgeon in charge of such lesions' removal (i) some actinic keratosis adjoining carcinoma to be resected therefore causing the problem of functional areas damaging (eyelids, lips, etc.) or (ii) numerous actinic keratosis localized away from carcinoma (photo-carcinogenesis field) faces the issue of clinical evaluation of such lesions: which ones will spontaneously regress (it is supposed to be the case for 20 % of such lesions);which ones will remain and which ones will develop into invasive carcinomas ?

A non-invasive, non-traumatic, automated and real-time help for the clinical diagnosis orientation of such skin lesions could help improving diagnosis accuracy of the medical practitioner's visual inspection:

* In terms of sensitivity in order to potentially decrease the number of actinic keratosis evolving towards invasive carcinoma,
* In terms of specificity in order to potentially decrease useless resections and reduce resection margins and therefore reduce scars surface.

ELIGIBILITY:
Inclusion Criteria:

* Adults, and
* Autonomous: enjoying full citizenship rights and full mental abilities, and
* Affiliated to a social security system, and
* Suffering from carcinomatous or polymorphous skin lesions that can be fully managed in an outpatient (ambulatory) surgery procedure.

Exclusion Criteria:

* Carcinomatous or polymorphous skin lesions that require day admission, or
* Carcinomatous or polymorphous skin lesions for which resection margins are uncertain, or
* Naevomatous skin lesions and related skin pathologies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-10; Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Optical spectroscopy's diagnostic validity for the 4 histological classes discrimination | day 1

SECONDARY OUTCOMES:
Statistical significance degree of the discrimination by molecular profiling (transcriptomic characterization) between in situ carcinoma (ISC) and invasive carcinoma (InvC). | day 1
Statistical significance degree of the discrimination by molecular profiling (transcriptomic characterization) between 2 classes of actinic keratosis (AK) of clinical relevance: AK characterized by a "low" versus a "high" invasiveness risk | day 1
- Sensitivity and specificity of optical spectroscopy for discriminating the é molecular classes of actinic keratosis: AK characterized by a "low" versus a "high" invasiveness risk. | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Khairallah, Principal Investigator — g.khairallah@chr-metz-thionville.fr
Locations (1):
- CHR Metz Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No